CLINICAL TRIAL: NCT01749488
Title: The Impact of Involving a Dietitian in the Implementation of Expert Recommendations Concerning Nutrition During Intensive Care on Energy Balance
Brief Title: The Impact of a Dietitian in the Implementation of Nutrition Recommendations During Intensive Care
Acronym: NutriSave
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The intervention becomes obsolete for participating centres pending regulatories.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRC-I/2012/SB-01; 2012-A00626-37 (Other: RCB number)
Record Dates: First submitted 2012-12-12; First posted 2012-12-13 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Intensive Care
Keywords: Dietitian; Nutritional recommendations; ICU nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control intensive care wards (No Intervention): This is a randomized cluster trial. The centers randomized into this arm will serve as controls. No interventions will be implemented for these centers.
- Experimental intensive care wards (Experimental): This is a randomized cluster trial. The centers randomized into this arm will designate a dietitian who will help the ward implement current recommendations for the nutrition of patients undergoing intensive care.
  Intervention: Designated dietitian for the ward
  Interventions: Other: Designated dietitian for the ward

INTERVENTIONS:
Other: Designated dietitian for the ward — This is a randomized cluster trial. The centers randomized into this arm will designate a dietitian who will help the ward implement current recommendations for the nutrition of patients undergoing intensive care.
  Arms: Experimental intensive care wards

SUMMARY:
The main objective of this study is to evaluate the impact of the intervention of a dietician on the energy balance accumulated over seven days of intensive care.

Energy balance is defined as the difference between the target recommended energy and total calorie intake actually received.

This is a randomized-cluster study; participating centers are randomized into experimental and control groups.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare the impact of the intervention of a dietician on:

* daily and accumulated energy balance at the end of the intensive care unit (ICU) stay
* deficits in protein intake per day, accumulated over 7 days, and accumulated for the ICU stay
* intake of vitamins, trace elements and pharmaco-nutrients per day
* predominant route of nutrition administration (enteral / parenteral / mixed)
* the course of the stay: duration of mechanical ventilation, organ failure, the ICU stay, number of days on antibiotics
* the presence / absence of complications: mortality, on catheter bacteremia, ventilator acquired pneumonia, other infections, bedsores, episodes of hyper-or hypoglycemia
* presence/absence of diarrhea
* costs related to the management of malnourished patients in terms of enteral and parenteral nutritional therapy, dietary supplements, antibiotics and sedatives as well as the costs of ICU stay and those related to diarrhea and sores

ELIGIBILITY:
Inclusion Criteria:

* The patient must be insured or beneficiary of a health insurance plan
* Patients hospitalized in intensive care for an expected period greater than 72 hours, and for whom sufficient eating after 72 hours of hospitalization is deemed unlikely upon admission.
* Patients receiving mechanical ventilation and having at least one organ failure other than respiratory failure, defined by a SOFA score greater than 2.

Exclusion Criteria:

* The patient is under judicial protection
* The patient (or his/her legal representative or "trusted-person") indicates they do not wish to participate in the study
* It is impossible to correctly inform either the patient or his/her "trusted person"
* The patient is participating in another study, or is in an exclusion period determined by another study
* Moribund patients or those for whom death appears imminent (within 24 hours)
* Survival to Day 28 unlikely due to uncontrollable comorbidities
* Patients with advanced directives issued expressing the wish to not be resuscitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Caloric deficit accumulated over 7 days | Day 7
  Caloric deficit accumulated over 7 days (kcal/kg)

SECONDARY OUTCOMES:
Average per day caloric deficit | Day 7
  Average per day caloric deficit (kcal/kg/day)
Caloric deficit accumulated during the ICU stay | ICU discharge (maximum of 28 days)
  Caloric deficit accumulated during the ICU stay (kcal/kg)
Average per-day protein deficit | Day 7
  Average per-day protein deficit (grams protein/kg/day)
Protein deficit accumulated over 7 days | Day 7
  Protein deficit accumulated over 7 days (grams protein/kg)
Protein deficit accumulated during the ICU stay | ICU discharge (maximum of 28 days)
  Protein deficit accumulated during the ICU stay (grams protein/kg)
Average per day amounts of vitamins received | Day 7
Average per day amounts of trace elements received | Day 7
Average per day amounts of pharmaco nutrients received | Day 7
Percentage of calories received by enteral route | Day 7
  daily average
Percentage of calories received by enteral route | Day 7
  accumulated over 7 days
Percentage of calories received by enteral route | ICU discharge (maximum of 28 days)
  accumulated over ICU stay
Percentage of proteins received by enteral route | Day 7
  daily average
Percentage of proteins received by enteral route | Day 7
  accumulated over 7 days
Percentage of proteins received by enteral route | ICU discharge (maximum of 28 days)
  accumulated over ICU stay
length of time spent on ventilator (hours) | ICU discharge (maximum of 28 days)
length of ICU stay (days) | ICU discharge (maximum of 28 days)
Number of days spent with (any) organ failure | ICU discharge (maximum of 28 days)
Number of days on antibiotics | ICU discharge (maximum of 28 days)
Mortality (yes/no) | Day 90
Mortality (yes/no) | Day 180
Presence/absence of on-catheter bacteremia | Day 7
Presence/absence of on-catheter bacteremia | Day 28
Presence/absence of on-catheter bacteremia | ICU discharge (maximum of 28 days)
Presence/absence of ventilator acquired pneumonia | Day 7
Presence/absence of ventilator acquired pneumonia | Day 28
Presence/absence of ventilator acquired pneumonia | ICU discharge (maximum of 28 days)
Presence/absence of other infections | Day 7
Presence/absence of other infections | Day 28
Presence/absence of other infections | ICU discharge (maximum of 28 days)
Presence/absence of bed sores | Day 7
Presence/absence of bed sores | Day 28
Presence/absence of bed sores | ICU discharge (maximum of 28 days)
Composite score for complications | Day 7
  Presence/absence of at least one of the following complications: on-catheter bacteremia, ventilator acquired pneumonia, other infections, bed sores
Composite score for complications | Day 28
  Presence/absence of at least one of the following complications: on-catheter bacteremia, ventilator acquired pneumonia, other infections, bed sores
Composite score for complications | ICU discharge (maximum of 28 days)
  Presence/absence of at least one of the following complications: on-catheter bacteremia, ventilator acquired pneumonia, other infections, bed sores
Minimum observed glycemia | Day 7
Minimum observed glycemia | ICU discharge (maximum of 28 days)
Maximum observed glycemia | Day 7
Maximum observed glycemia | ICU discharge (maximum of 28 days)
Average observed glycemia | Day 7
Average observed glycemia | ICU discharge (maximum of 28 days)
Presence/absence of a glycemia measure < 0.4 g/l | Day 7
Presence/absence of a glycemia measure < 0.4 g/l | ICU discharge (maximum of 28 days)
Presence/absence of a glycemia measure > 1.8 g/l | Day 7
Presence/absence of a glycemia measure > 1.8 g/l | ICU discharge (maximum of 28 days)
Presence/absence of hypertriglyceridemia | Day 7
Presence/absence of hypertriglyceridemia | ICU discharge (maximum of 28 days)
Accumulated cost of enteral nutrition | Between Day 0 and ICU discharge (expected maximum of 28 days)
Accumulated cost of parenteral nutrition | Between Day 0 and ICU discharge (expected maximum of 28 days)
Accumulated cost of antibiotics | Between Day 0 and ICU discharge (expected maximum of 28 days)
Accumulated cost of sedation | Between Day 0 and ICU discharge (expected maximum of 28 days)
Presence/absence of diarrhea | Between Day 0 and ICU discharge (expected maximum of 28 days)
Accumulated cost of nutritional supplements | Between Day 0 and ICU discharge (expected maximum of 28 days)
Accumulated cost of ICU stay | Between Day 0 and ICU discharge (expected maximum of 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Saber Davide Barbar, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes; Jean-Yves Lefrant, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes